CLINICAL TRIAL: NCT06385340
Title: Investigation of the Effect of Lipikar Baume AP+M on Skin Barrier, Microbiome and AKASI of Participants With Actinic Keratoses and Field Cancerization of the Forearms and Hands
Brief Title: Investigation of the Effect of Lipikar Baume AP+M
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CentroDerm GmbH (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CentroDerm_LRP22003
Record Dates: First submitted 2024-04-02; First posted 2024-04-26 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Actinic Keratoses
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Intervention Model Description: It's a randomized, evaluator blinded, intra-individual controlled study conducted in one center in Germany, in adult subjects having AK (grade I to III) lesions on the forearms and back of hands and meeting specific inclusion/exclusion criteria.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lipikar Baume AP+M (Other): Application of Lipikar Baume AP+M at least twice daily for 4 weeks on one of the two arms according to a randomization scheme
  Interventions: Other: Lipikar Baume AP+M
- no intervention (No Intervention): Application of Lipikar Baume AP+M at least twice daily for 4 weeks on one of the two arms according to a randomization scheme

INTERVENTIONS:
Other: Lipikar Baume AP+M — • Lipikar Baume AP+M Application of Lipikar Baume AP+M at least twice daily for 4 weeks on one of the two arms according to a randomization scheme
  Arms: Lipikar Baume AP+M

SUMMARY:
Application of Lipikar Baume AP+M at least twice daily for 4 weeks on one of the two arms according to a randomization scheme The purpose of this study is to observe the skin barrier function, transepidermal water loss and microbial changes in study participants with actinic field damage of both arms.

It's a randomized, evaluator blinded, intra-individual controlled study conducted in one center in Germany, in adult subjects having AK (grade I to III) lesions on the forearms and back of hands and meeting specific inclusion/exclusion criteria.

A total of 20 subjects will be enrolled.

The study design consists in 4-week evaluation period, with 2 visits per subject: Screening/Baseline (Day 0, Day 28 (end of Lipikar Baume AP+M application)).

ELIGIBILITY:
Inclusion Criteria:

* Male, female, diverse persons (> 18yo) who are capable of giving consent
* Female patients are eligible if the subject is not a woman of childbearing potential (WOCBP) or if she is postmenopausal (cessation of menstruation >12 months) or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, total hysterectomy)
* Signed informed consent
* Diagnosis of at least 4 actinic keratoses of the the forearm and/or back of the hand (each arm)
* Olsen grade I, II and/or III
* Subjects with similar severity and number of AKs on each side symmetrically
* The study participant is in good general condition for his or her age and does not currently have any active diseases that, in the opinion of the investigator, justify exclusion from the study

Exclusion Criteria:

* Known or documented intolerance to any of the ingredients of Lipikar Baume AP+M
* Any planned AK treatment during the study
* Treatment of actinic keratoses in the application area within the past 3 Months (e.g. photodynamic therapy, topical 5-FU, diclofenac, imiquimod, cryotherapy etc.)
* Suspected invasive squamous cell cancer in the application area
* Chronic wounds, erosions, pre-existing infected skin or inflammation which, in the opinion of the investigator, are in need of treatment other than the study product
* Suspected non-compliance
* Current or within the last 8 weeks given systemic cancer medication or systemic treatment with 5-Fluorouracil
* Any systemic immunosuppressant given within the 8 weeks prior to the study (e.g. systemic prednisolone, azathioprine etc.)
* Locally applied retinoids, steroids, or other prescribed externals in the 4 weeks prior to the start of the study that, in the opinion of the study physician, necessitate exclusion
* Products containing glycolic or alpha-hydroxy acids applied locally in the application area in the last 4 weeks
* Participation in another clinical trial
* Participation in a clinical study within the last 30 days
* Family members or colleagues of the investigator
* Participant is in a position or has a relationship with the investigator that presents a potential conflict of interest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-23 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Skin hydration measured by Corneometrie | Day 28
  Corneometer® (Courage + Khazaka electronics GmbH, Cologne, Germany) is used to assess skin hydration after 28 days. The Corneometer® measures in arbitrary units from 0 (no water) - 120 (on water). The units are referred to as "Corneometer® units". In total there will be 3 measurements at each point (Actinic keratosis, perilesional, never by actinic keratosis affected skin/healthy). The average of the 3 measurements is calculated and day 0 and day 28 are compared.
Transepidermal water loss measured by Tewameter® | Day 28
  Transepidermal water loss (in g/m2/h - TEWL) measured by Tewameter® (Courage + Khazaka electronics GmbH, Cologne, Germany). 3 measurements at each arm und lesion will be taken (Actinic keratosis, perilesional and never by actinic keratosis affected skin). The average of the 3 measurements is calculated and day 0 and day 28 are compared.
Aktinic keratosis area and severity index (AKASI) | Day 28
  The AKASI is a standardized tool for the clinically adequate assessment of larger areas (1). The area, distribution, erythema, and thickening of actinic keratoses are evaluated according to Dirschka et al. and a score is calculated. The score is between 0-18. Average values of study participants of each study group will be compared (day 0, day 28).
  1. Dirschka T, Pellacani G, Micali G, Malvehy J, Stratigos AJ, Casari A, et al. A proposed scoring system for assessing the severity of actinic keratosis on the head: actinic keratosis area and severity index. J Eur Acad Dermatol Venereol. 2017;31(8):1295-302.
S. aureus colonization and S. epidermidis colonization (application area) | Day 28
  S. aureus colonization and S. epidermidis colonization is assessed after 28 days by skin swabs and qPCR. Quantification is based on fluorescence measurements taken in real time during a PCR cycle. Fluorescence increases in proportion to the amount of PCR product. At the end of a run (consisting of several cycles), quantification is performed in the exponential phase of the PCR using the fluorescence signals obtained. Mean Ct values (cycle threshold) of the study groups are given for qPCR.
Subjects's skin aspect | Day 28
  The investigator will assess the subject's skin aspect on the following signs or symptoms: scarring, atrophy, induration, redness or change in pigmentation.
  The Score is between 0 (poor) and 3 (Excellent). The investigator will assess the subjects skin aspect at day 28 for all lesions, that have disappeared. An anverage of the score is calculated for all lesions in each study group.

SECONDARY OUTCOMES:
Absolute lesion count by application site | Day 28
  Actinic keratoses that are clearly visible or palpably are counted at each study site (left and right arm and back of the hands).
  Absolute lesion counts by application site will be compared (day 0 and day28).
Olsen Grade evaluation: percentage of lesion with improvement at least 1 grade at D28 by application site | Day 28
  The percentage of lesions with an improvement of at least one grade (Olsen grade) at day 28 will be assessed.
  For this the Olsen classification of each actinic keratosis should be recorded. This classification is based on a three-grade grading of the thickness of a single lesion and was first proposed by Olsen et al. Grade 1 describes a slightly palpable lesion, grade 2 a moderately thick and grade 3 a very thick and hyperkeratotic lesion. If actinic field cancerization is present, the highest Olsen grade in the area will be assessed.
  Average Olsen Scores by application site of Day 0 and D28 will be compared.
Number of new lesions on application area over the study period by application site | Day 28
  All new actinic keratoses in the study area are recorded by application site (left and right arm and back of the hands).
  Day 0 and Day 28 will be compared concerning the average of new lesions by application site.
Symptom severity score: percentage across individual scores at each visit by application site | Day 28
  A symptom score with a four-point Likert scale (absent, light, moderate, severe) is assessed as patient reported outcome (PRO). The symptom score includes four principal symptoms (itch, unpleasant burning, pain, tingling).
  The paper questionnaire with 4 questions will be handed out to the patient at Day 0 and Day 28. The symptom score is assessed for botch arms separately. The average scores by application will be compared concerning the overall score and the individual symptom scores (itch, burning etc.) at day 0 and day 28.
modified Treatment Satisfaction Questionnaire for Medication-9 (mTSQM-9) | Day 28
  To assess the general satisfaction with Lipikar Baume AP+M an according to the study procedures modified TSQM-9 will be applied. This is a questionnaire that has been evaluated for the evaluation of antihypertensive medications but can also be applied to dermatological diseases.
  This includes nine questions with Likert-scaled answers to assess the satisfaction with the cosmetic.
  As the TSQM-9 was developped for medical agents, we changed the word medicament to "cosmetic", to assess the score at day 0 and day 28. The average of score of day 0 and day 28 will be compared.
Compliance (percentage of subjects using topical agents at all intended days, 90% of days or 75% of days) | Day 28
  A patient diary is used to assess the days on which Lipikar Baume AP+M was used.
  The proportion of patients with at least 75% of days and >90% of days on which Lipikar Baume AP+M was used will be calculated.
Pictures at all time points | Day 28
  Pictures of the forearms and back of the hands are taken to illustrate the effects of Lipikar Baume AP+M.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Dirschka, Prof. Dr., Principal Investigator — CentroDerm GmbH
Locations (1):
- CentroDerm GmbH, Wuppertal, North Rhine-Westphalia, Germany